CLINICAL TRIAL: NCT02171663
Title: A Phase I Open-label Dose Escalation Study of Once-daily Oral Treatment With BIBF 2992 for 21 Days in Patients With Advanced Solid Tumors
Brief Title: Dose Escalation Study of BIBW 2992 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.2
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib

ARMS (1):
- BIBW 2992 (Experimental)
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992

SUMMARY:
The primary objective was the assessment of safety of BIBW 2992 as assessed by the maximum tolerated dose (MTD). Secondary objectives were collection of overall safety data, antitumor efficacy data, as well as the determination of pharmacokinetics and the pharmacodynamic modulation of biomarkers by BIBW 2992.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with confirmed diagnosis of advanced, non resectable and / or metastatic solid tumors, of types historically known to express EGFR and/or HER2, who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment preferably patients with breast, colorectal or prostate cancer
* Age 18 years or older
* Life expectancy of at least three (3) months
* Written informed consent given that is consistent with International Conference on Harmonization - Good Clinical Practice guidelines
* Eastern Cooperative Oncology Group (ECOG) performance score 0, 1, or 2
* Patients must have resolution of prior chemo-, hormone, immuno-, or radiotherapy-related toxicities to CTC Grade <= 1 or baseline
* Patients have to be recovered from previous surgery

The 12 additional patients recruited at the MTD must also meet the following criteria:

* Measurable tumor deposits (RECIST) by one or more techniques (X-ray, CT, MRI)

Exclusion Criteria:

* Active infectious disease
* Gastrointestinal disorders that might interfere with the absorption of the study drug or chronic diarrhea
* Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
* Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least eight weeks, no history of cerebral edema or bleeding in the past eight weeks and no requirement for steroids or anti-epileptic therapy
* Cardiac left ventricular function with resting ejection fraction ≥ CTC Grade 1
* Absolute neutrophil count (ANC) less than 1500 / mm3
* Platelet count less than 100 000 / mm3
* Bilirubin greater than 1.5 mg / dl (> 26 μmol / L, SI unit equivalent)
* Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than three times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
* Serum creatinine greater than 1.5 mg / dl (> 132 μmol / L, SI (Système Internationale) unit equivalent)
* Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
* Pregnancy or breast-feeding
* Treatment with other investigational drugs; chemotherapy, immunotherapy, radiotherapy or hormone therapy (excluding Luteinizing Hormone-Releasing Hormone agonists, other hormones taken for breast cancer, or bisphosphonates) or participation in another clinical study within the past four weeks before start of therapy or concomitantly with this study
* Treatment with an EGFR- or HER2 inhibiting drug within the past four weeks before start of therapy or concomitantly with this study (8 weeks for trastuzumab)
* Patients unable to comply with the protocol
* Active alcohol or drug abuse

The patient may be eligible for re-treatment after the previous course finished. The patient will not be eligible if the following criteria are met:

* Patients with clinical signs of disease progression or if latest X-ray, CT or MRI reveals progressive disease
* Cardiac left ventricular function CTC Grade ≥ 2 at any time during the previous course
* Patients fulfilling any of the Exclusion Criteria as mentioned before on Day 29 of the previous course
* Patients not recovered from any dose-limiting toxicity (DLT) 14 days after the last administration of BIBW 2992 in the previous course. Recovery is defined as a return to baseline level or CTC Grade 1, whichever is higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-03; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | up to 22 months
Incidence and intensity of Adverse Events (AE) according to Common Terminology Criteria (CTC Version 3), that were associated with increasing doses of BIBW 2992 | up to 22 months

SECONDARY OUTCOMES:
Assessment of biomarker modulation (EGFR, p-EGFR, p-MAPK (mitogen-activated protein kinase), p-Akt, Ki 67, p-27KIP1) in skin biopsies | Baseline and day 21 of the first treatment period
Assessment of biomarker modulation (EGFR, p-EGFR, Her2, p-MAPK, p-Akt, Ki 67, p-27KIP1) in tumor biopsies in six or more patients treated at the MTD | Baseline and day 21 of the first treatment period
Objective tumor responses | up to 22 months
Correlation of EGFR, HER2, estrogen receptor (ER) and progesterone receptor (PrR) immunohistochemical status, based on tumor biopsies or excisions obtained prior to this trial, with objective tumor responses | up to 22 months
Area under the plasma concentration time curve (AUC) for different time points | up to 72 hours after last dose on day 21
Percentage of AUC0-infinity that is obtained by extrapolation (%AUC0-tz) | up to 72 hours after last dose on day 21
Predose plasma concentration (Cpre) for different time points | Day 8, 15 and 21
Plasma concentration (C) | 24 hours after the first dose on day 1 and the last dose on day 21
Maximum measured plasma concentration (Cmax) for different time points | up to 72 hours after last dose on day 21
Time from dosing to the maximum plasma concentration (tmax) for different time points | up to 72 hours after last dose on day 21
Terminal half-life (t1/2) for different time points | up to 72 hours after last dose on day 21
Mean residence time after oral administration (MRTpo) for different time points | up to 72 hours after last dose on day 21
Apparent clearance (CL/F) for different time points | up to 72 hours after last dose on day 21
Apparent volume of distribution during the terminal phase (Vz/F) for different time points | up to 72 hours after last dose on day 21
Accumulation ratio (RA) with respect to Cmax and AUC | up to 72 hours after last dose on day 21